CLINICAL TRIAL: NCT06291181
Title: Studying the Distribution of Accessory Gene Regulator (Agr) Quorum Sensing System and the Prevalence of Linezolid and Mupirocin Resistance in Biofilm Producer/Non Producer Staphylococcus Aureus in Sohag University Hospitals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Bakry, assistant specialist at fever hospital, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Soh-Med-24-01-05MD
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Staphylococcus Aureus
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cases group (Experimental): wound infected patients
  Interventions: Diagnostic Test: antibiotic sensitivity test

INTERVENTIONS:
Diagnostic Test: antibiotic sensitivity test — Disc diffusion method using modified Kirby-Bauer technique on Muller Hinton agar (MHA) will be carried out for antimicrobial susceptibility of S. aureus isolates. The following antibiotics will be tested: cefoxitin (30 µg ), Tetracyclin 30 µg (TE), Chloramphenicol 30 µg (C), Gentamycin 10µg (CN), Erythromycin 15µg(E),Clindamycin 2 µg (DA), Ciprofloxacin 5 µg (CIP), Trimethoprim/sulphamethoxazole 1.25/23.75 µg (SXT), Rifampin 5µg (RA), Linezolide 30µg (LZD); cefoxitin disc (FOX 30 g)
  zone diameters interpretation will be done according to Clinical and Laboratory Standard Institute (CLSI 2018),

SUMMARY:
Staphylococcus aureus is an important pathogen causing a wide spectrum of infections . The organism usually colonizes the skin and mucous of humans and several animal species. Multiple body sites can be colonized in humans, however, the anterior nares of the nose are the most frequent carriage site for S. aureus. Other sites for carriage include the skin, perineum, and pharynx . It has been shown that there is an increased prevalence of staphylococcus infections, which may be attributed to its carriage in anterior nares and hands of health care workers and patients .

The pathogenic mechanisms enabling S. aureus to cause serious infections could include: biofilm which protects organisms from host immune response; opsonophagocytosis and antimicrobial agents, thus leading to chronic and persistent infections.

Antibiotic resistance associated with S.aureus infections is a great concern for the clinicians to prevent spread of infections. Methicillin was commonly used for these infections before the emergence of MRSA which is developed due to irrational use of antibiotics, prolonged hospital stay, nasal and hand carriage in health care staff. Also vancomycin, linezolid and mupirocin are used in treating infections,as well as decolonization of carriers .

Mupirocin act by inhibiting the protein synthesis of bacteria by binding specifically to isoleucyl-tRNAsynthetase enzyme. The irrational use of Mupirocin among patients and its carriage in health care staff has led to the emergence of resistance to this antibiotic. .

MupA, plasmid mediated gene, has a great role in mupirocinresistence as it had a supplementary modified isoleucyltRNAsynthetase which leads to the high level resistance to Mupirocin. The mupA gene has the ability to facilitate and disseminate the resistance mechanism in different patterns .

Linezolid,theﬁrstoxazolidinonedrug,waslaunchedin2001andis still displaying excellent in vitro activity against Staphylococcus epidermidis on a global scale,although outbreaks of linezolidresistant S. epidermidis (LRSE) are occasionally reported..

Linezolid resistance is mediated by, mutations in the 23S rRNA gene, altering the drug-binding site, and/or the 50S ribosomal proteins L3, L4 and L22, impairing linezolid binding;,Oracquisition of the primarily plasmid-encoded genes cfr, encoding a methyltransferase, or optrA, encoding an ABC transporter, or the cfr homologues cfr(B) and cfr(C).

While cfr can mediate the PhLOPSA phenotype (resistance to phenicols, lincosamides,oxazolidinones, pleuromutilins and streptogramin A compounds), optrA confers oxazolidinone and phenicolresistance only..

Pathogenecity of S. aureus is regulated by various factors ,one of them is the accessory gene regulatory (agr) system. It consists of 2 divergently transcribed loci (3 kb) controlled by means of 2 promoters P2 and P3. Most of clinical isolates of acute infections have a functional agr system and all, like strains, produce RNAIII in vitro and in vivo.

Agr deficiency has been related to increased biofilm formation because RNAIII reduces the expression of surface adhesins and increases the production of capsule, toxins, and proteases. The agr system is supposed to regulate over 70 genes, 23 of which are renowned virulence factors.

There are 2 classes of virulence factors regulated by agr. The first class includes virulence factors implicated in attachment to the host and immune evasion, whereas the second class contains genes engaged in the production of exoproteins related to invasion and toxin production . The activation of the agr system switches the bacterium from an adhesive, colonizing commensal into an invasive and aggressive pathogen(Roux A et al; 2009).

Major virulence factors in S. aureus, exfoliative toxins (ETs), toxic shock syndrome toxin (TSST-1), and staphylococcal enterotoxins (SEs) are involved in host colonization, invasion of damaged skin and mucus, gastrointestinal infection, and prevarication of host defense mechanisms. Indeed, agr operon including agrA, agrB, agrC, and agrD genes regulate over 70 genes in S. aureus 23 of which control its pathogenicity and invasive infections .

Moreover, S. aureus can be stratified into 4 different groups (agr I, agr II, agr III, and agr IV) according to the sequences of agrC (auto inducing peptide) and agrD (cyclic AIP) genes. It is stated that agr types are different in their properties and prevalence in various geographical areas thus, identification of predominant types in each region may well be functional .

ELIGIBILITY:
Inclusion Criteria:

* patients with signs of wound infection like pus or exudate

Exclusion Criteria:

* burns with greenish discharge and wounds with fungal infection

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
resistence of staphylococci to mupirocin and linezolid antibiotics | 6 months
  Antibiotic resistance associated with S.aureus infections is a great concern for the clinicians to prevent spread of infections. .
  Mupirocin act by inhibiting the protein synthesis of bacteria by binding specifically to isoleucyl-tRNAsynthetase enzyme. The irrational use of Mupirocin among patients and its carriage in health care staff has led to the emergence of resistance to this antibiotic..
  Linezolid resistance is mediated by, mutations in the 23S rRNA gene, altering the drug-binding site, and/or the 50S ribosomal proteins L3, L4 and L22, impairing linezolid binding;),Oracquisition of the primarily plasmid-encoded genes cfr, encoding a methyltransferase, or optrA, encoding an ABC transporter, or the cfr homologues cfr(B) and cfr(C).

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Anderson DJ, Kaye KS. Staphylococcal surgical site infections. Infect Dis Clin North Am. 2009 Mar;23(1):53-72. doi: 10.1016/j.idc.2008.10.004. PMID 19135916
- [Background] Anderson DJ, Podgorny K, Berrios-Torres SI, Bratzler DW, Dellinger EP, Greene L, Nyquist AC, Saiman L, Yokoe DS, Maragakis LL, Kaye KS. Strategies to prevent surgical site infections in acute care hospitals: 2014 update. Infect Control Hosp Epidemiol. 2014 Sep;35 Suppl 2:S66-88. doi: 10.1017/s0899823x00193869. No abstract available. PMID 25376070
- [Background] Arciola CR, Baldassarri L, Montanaro L. Presence of icaA and icaD genes and slime production in a collection of staphylococcal strains from catheter-associated infections. J Clin Microbiol. 2001 Jun;39(6):2151-6. doi: 10.1128/JCM.39.6.2151-2156.2001. PMID 11376050